CLINICAL TRIAL: NCT04466124
Title: Prospective Cohort Study for Identifying Factors Predicting Clinical Outcomes of Liver Cancer Patients Treated With Proton Beam Therapy
Brief Title: Prospective Cohort Study of Liver Cancer Patients Treated With Proton Beam Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC2018-0197
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Liver Cancer
Keywords: Proton Beam Therapy; Cohort Study
MeSH Terms: conditions — Liver Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Liver Cancer Patients Treated With Proton Beam Therapy — Proton Beam Therapy

SUMMARY:
Liver cancer is the fourth most common malignant tumor in Korea and it is the third most common cause of cancer death worldwide according to the 2009 Korea Central Cancer Registration Annual Report. Excellent survival rate (50-70% 5-year survival rate) can be obtained when surgery is performed including liver transplantation, but most (70-80%) patients with liver cancer are difficult to get surgery due to liver disease associated with cirrhosis. In addition, due to the multi-centric nature of liver cancer in patients with cirrhosis, repeated treatment is required. For these reasons, various treatments for liver cancer (percutaneous arterial embolization, percutaneous ethanol injection, radiofrequency heat therapy, and radiation therapy) have been performed.

Due to recent advances in radiotherapy technology, proton beam therapy (PBT) is a promising treatment for liver cancer because it maximizes radiation to tumor tissues and reduces radiation doses from surrounding normal tissues due to the distinct physical properties of proton beams. Promising therapeutic results and less toxicity have been reported in liver cancer. In addition, several genes in liver cancer (SOCS-1, GSTP, APC, VEGF, PD-EGF, HIF-1, NOS, b-FGF, LINE-1, p27, TOP2A, Ets-1, Bcl-xL, Osteopontin, CD44, etc.) have been reported to be associated with recurrence and prognosis.

DETAILED DESCRIPTION:
Liver cancer is the fourth most common malignant tumor in Korea and it is the third most common cause of cancer death worldwide according to the 2009 Korea Central Cancer Registration Annual Report. Excellent survival rate (50-70% 5-year survival rate) can be obtained when surgery is performed including liver transplantation, but most (70-80%) patients with liver cancer are difficult to get surgery due to liver disease associated with cirrhosis. In addition, due to the multi-centric nature of liver cancer in patients with cirrhosis, repeated treatment is required. For these reasons, various treatments for liver cancer (percutaneous arterial embolization, percutaneous ethanol injection, radiofrequency heat therapy, and radiation therapy) have been performed.

Due to recent advances in radiotherapy technology, proton beam therapy (PBT) is a promising treatment for liver cancer because it maximizes radiation to tumor tissues and reduces radiation doses from surrounding normal tissues due to the distinct physical properties of proton beams. Promising therapeutic results and less toxicity have been reported in liver cancer. In addition, several genes in liver cancer (SOCS-1, GSTP, APC, VEGF, PD-EGF, HIF-1, NOS, b-FGF, LINE-1, p27, TOP2A, Ets-1, Bcl-xL, Osteopontin, CD44, etc.) have been reported to be associated with recurrence and prognosis. Therefore, in this study, the investigator is going to establish a prospective cohort of liver cancer patients treated with proton beam therapy. It be used for analyzing local control, survival, recurrence, toxicity, proton treatment plan information, gene expression information, then local control (LC), overall survival. (overall survival, OS), recurrence-free surival (RFS), and factors that predict treatment-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer patients scheduled to be proton beam therapy
* Agreed to participate in this study

Exclusion Criteria:

-Disagreed to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver cancer patients over the age of 19
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Establish a cohort of liver cancer patients treadted with proton beam therapy. | Up to 10 years
  The primary outcome is to establish a prospective cohort of liver cancer patients treadted with proton beam therapy. It is for exploration of factors and models that predict local control, recurrence, survival and treatment-related toxicity in liver cancer patients undergoing proton therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hyun Kim, Ph.D, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea